CLINICAL TRIAL: NCT00812461
Title: Nalmefene Efficacy Study II: Randomised, Double-blind, Placebo-controlled, Parallel-group, Efficacy Study of 20 mg Nalmefene, as Needed Use, in Patients With Alcohol Dependence
Brief Title: Efficacy of Nalmefene in Patients With Alcohol Dependence
Acronym: ESENSE2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12023A; 2007-002563-27 (EudraCT Number)
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Alcohol Dependence
Keywords: Pharmacologic Actions; Alcohol-Related Disorders; Alcoholism; Mental Disorders; Central Nervous System Agents
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Mental Disorders | interventions — nalmefene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Nalmefene (Experimental)
  Interventions: Drug: Nalmefene

INTERVENTIONS:
Drug: Placebo — as-needed use, tablets, orally, 6 months
  Arms: Placebo
Drug: Nalmefene — 18.06 mg, as-needed use, tablets, orally, 6 months. 18.06 mg nalmefene equals 20 mg nalmefene hydrochloride.
  Other Names: Selincro™
  Arms: Nalmefene

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety and tolerability of nalmefene in the treatment of alcohol dependence.

DETAILED DESCRIPTION:
Alcohol dependence is a maladaptive pattern of alcohol use, leading to clinically significant impairment or distress, as manifested by at least three of a number of criteria such as tolerance, withdrawal symptoms, frequent use of alcohol in larger amounts or over longer periods than was intended, and others. Excessive intake of alcohol reduces the life span by a decade, and alcohol drinking is strongly related to mortality from liver cirrhosis, chronic pancreatitis, certain cancers, hypertension, accidents and violence. This study is planned to evaluate the efficacy and safety of as needed use of nalmefene 18.06 mg versus placebo in decreasing monthly Heavy Drinking Days (HDDs) and decreasing the total consumption during a period of 24 weeks in adult patients with alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

In- and outpatients who:

* had a primary diagnosis of alcohol dependence according to Diagnostic and Statistical Manual of Mental Disorders - text revision (DSM-IV-TR) criteria
* had had ≥6 HDDs in the 4 weeks preceding the Screening Visit
* had had an average alcohol consumption at WHO medium risk level or above in the 4 weeks preceding the Screening Visit

Exclusion Criteria:

The patient:

* had a DSM-IV Axis I disorder other than alcohol dependence or nicotine dependence
* had an antisocial personality disorder
* had risk of suicide evaluated by the suicidality module of the Mini-International Neuropsychiatric Interview (MINI)
* had a history of delirium tremens or alcohol withdrawal seizures
* reported current or recent (within 3 months preceding screening) treatment with disulfiram, acamprosate, topiramate, naltrexone or carbimide, or with any opioid antagonists
* reported current or recent treatment with antipsychotics or antidepressants
* was pregnant or breast-feeding

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (57):
- Belgium (7):
  - BE002, Assebroek
  - BE007, Bruges
  - BE006, Charleroi
  - BE005, Kortenberg
  - BE001, Liège
  - BE003, Mechelen
  - BE004, Ostend
- Czechia (3):
  - CZ001, Litoměřice
  - CZ002, Prague
  - CZ003, Prague
- France (16):
  - FR008, Angers
  - FR004, Bully-les-Mines
  - FR009, Clichy
  - FR012, Élancourt
  - FR021, La Rochelle
  - FR011, Le Pecq
  - FR019, Lille
  - FR016, Lyon
  - FR014, Nancy
  - FR015, Nîmes
  - FR002, Rennes
  - FR001, Sartrouville
  - FR007, Strasbourg
  - FR005, Toulouse
  - FR006, Toulouse
  - FR003, Villejuif
- Italy (10):
  - IT017, Bologna
  - IT013, Bologna
  - IT008, Cento
  - IT006, Florence
  - IT002, Parma
  - IT007, Rome
  - IT001, Rome
  - IT011, Rome
  - IT004, Rome
  - IT018, Soverato Marina
- Poland (7):
  - PL005, Gdansk
  - PL004, Leszno
  - PL006, Lublin
  - PL007, Lublin
  - PL002, Piekary Śląskie
  - PL003, Skorzewo
  - PL001, Szczecin
- Portugal (4):
  - PT003, Angra do Heroísmo
  - PT002, Lisbon
  - PT001, Lisbon
  - PT006, Mem Martins
- Spain (10):
  - ES005, Alicante
  - ES006, Barcelona
  - ES008, Barcelona
  - ES004, Barcelona
  - ES014, Burgos
  - ES010, Madrid
  - ES001, Mallorca
  - ES002, Oviedo
  - ES003, Valencia
  - ES011, Zamora

REFERENCES:
- [Result] Gual A, He Y, Torup L, van den Brink W, Mann K; ESENSE 2 Study Group. A randomised, double-blind, placebo-controlled, efficacy study of nalmefene, as-needed use, in patients with alcohol dependence. Eur Neuropsychopharmacol. 2013 Nov;23(11):1432-42. doi: 10.1016/j.euroneuro.2013.02.006. Epub 2013 Apr 3. PMID 23562264
- [Derived] Aubin HJ, Reimer J, Nutt DJ, Bladstrom A, Torup L, Francois C, Chick J. Clinical relevance of as-needed treatment with nalmefene in alcohol-dependent patients. Eur Addict Res. 2015;21(3):160-168. doi: 10.1159/000371547. Epub 2015 Mar 31. PMID 25832297
- [Derived] Laramee P, Brodtkorb TH, Rahhali N, Knight C, Barbosa C, Francois C, Toumi M, Daeppen JB, Rehm J. The cost-effectiveness and public health benefit of nalmefene added to psychosocial support for the reduction of alcohol consumption in alcohol-dependent patients with high/very high drinking risk levels: a Markov model. BMJ Open. 2014 Sep 16;4(9):e005376. doi: 10.1136/bmjopen-2014-005376. PMID 25227627
- [Derived] van den Brink W, Aubin HJ, Bladstrom A, Torup L, Gual A, Mann K. Efficacy of as-needed nalmefene in alcohol-dependent patients with at least a high drinking risk level: results from a subgroup analysis of two randomized controlled 6-month studies. Alcohol Alcohol. 2013 Sep-Oct;48(5):570-8. doi: 10.1093/alcalc/agt061. Epub 2013 Jul 19. PMID 23873853

RESULTS

PARTICIPANT FLOW:
Groups:
- Nalmefene 18.06 mg: as-needed use, tablets, orally, 6 months
Period: All Randomised Patients
Arm/Group | Placebo | Nalmefene 18.06 mg
Started | 360 | 358
Completed | 337 | 341
Not Completed | 23 | 17
Not completed — Did not receive placebo/nalmefene | 23 | 17
Period: All Treated Patients
Arm/Group | Placebo | Nalmefene 18.06 mg
Started | 337 | 341
Completed | 205 (Patients who had the final visit of the study protocol) | 194 (Patients who had the final visit of the study protocol)
Not Completed | 132 | 147
Not completed — Adverse Event | 8 | 15
Not completed — Lack of Efficacy | 13 | 7
Not completed — Non-compliance | 6 | 9
Not completed — Protocol Violation | 36 | 27
Not completed — Withdrawal by Subject | 45 | 54
Not completed — Lost to Follow-up | 11 | 14
Not completed — Other Reason | 13 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nalmefene 18.06 mg | Total
Number analyzed (Participants) | 360 | 358 | 718
Age Continuous [Mean (Standard Deviation); unit: years] — All-patients-randomised set (APRS).
  years | 44.4 (10.7) | 45.1 (10.7) | 44.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants] — APRS.
  Participants
    Female | 104 | 92 | 196
    Male | 256 | 266 | 522
Previously Treated for Alcohol Dependence [Number; unit: participants] — APRS
  participants
    NO | 213 | 215 | 428
    YES | 147 | 142 | 289
    UNKNOWN | 0 | 1 | 1
Previously Treated for Alcohol Withdrawal Symptoms] [Number; unit: participants] — APRS.
  participants
    NO | 292 | 300 | 592
    YES | 68 | 57 | 125
    UNKNOWN | 0 | 1 | 1
Total Monthly Heavy Drinking Days (HDD) [Mean (Standard Deviation); unit: days] — APRS.
  Based on Timeline Followback (TLFB) data from the month preceding the screening visit.
  days | 18.37 (7.03) | 19.71 (6.96) | 19.04 (7.03)
Total Alcohol Consumption (TAC) g Alcohol/Day [Mean (Standard Deviation); unit: g] — APRS.
  Based on TLFB data from the month preceding the screening visit.
  g | 88.76 (48.15) | 92.22 (46.87) | 90.49 (47.52)
Drinking Risk Level (DRL) [Number; unit: participants] — APRS.
  participants
    Low | 6 | 5 | 11
    Medium | 82 | 68 | 150
    High | 134 | 129 | 263
    Very High | 138 | 156 | 294
Clinical Global Impression - Severity of Illness (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — APRS.
  The Clinical Global Impression - Severity of Illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 3.99 (1.42) | 4.05 (1.45) | 4.02 (1.44)
Gamma-glutamyl Transferase (GGT) [Mean (Standard Deviation); unit: international units per liter (IU/L)] — APRS.
  international units per liter (IU/L) | 97.39 (165.12) | 91.98 (153.01) | 94.69 (159.09)
Alanine Aminotransferase (ALAT) [Mean (Standard Deviation); unit: IU/L] — APRS.
  IU/L | 34.32 (26.06) | 34.20 (22.70) | 34.26 (24.42)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Monthly Number of Heavy Drinking Days (HDDs)
Description: Number of HDDs over a month (28 days), where one HDD was defined as a day with alcohol consumption ≥60 grams (g) for men and ≥40 g for women.
Time Frame: Baseline and Month 6
Population: Full-analysis set (FAS) - all patients in the all-patients-treated set (APTS) who had at least one valid post-baseline assessment in the main treatment period of both co-primary efficacy variables (HDD and TAC) and had an average alcohol consumption at medium Drinking Risk Level (DRL) or above according to WHO criteria at Baseline.
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 229 | 212
days | -10.58 (0.52) | -12.30 (0.54)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; The primary hypothesis concerned the treatment effect at Month 6. The null hypothesis of no difference in treatment effect was tested against the alternative hypothesis that there was a difference in treatment effect. MMRM model with the Baseline score as a covariate; site, sex, time in months (Month 1-6); and treatment as fixed effects. The Baseline score-by-time and treatment-by-time interactions were also included in the model. An unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.012, Adjusted change from Baseline to Month 6; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-3.07 to -0.38], Standard Error of Mean 0.68 — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 229 participants in the placebo group and 212 participants in the nalmefene group

2. Primary Outcome: Change From Baseline in the Monthly Total Alcohol Consumption (TAC)
Description: TAC was defined as mean daily alcohol consumption in g/day over a month (28 days).
Time Frame: Baseline and Month 6
Population: FAS
Measure: Mean (Standard Error); unit: g
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 229 | 212
g | -54.06 (2.23) | -59.01 (2.29)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.088, Adjusted change from Baseline to Month 6; Mean Difference (Final Values) = -4.95, 95% CI 2-sided [-10.63 to 0.73], Standard Error of Mean 2.89 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Drinking Risk Level (RSDRL) Response
Description: RSDRL response was defined as a downward shift from baseline in Drinking Risk Level (DRL); for patients at very high risk at Baseline: a shift to medium risk or below, and for patients at high or medium risk at Baseline: a shift to low risk or below.
Time Frame: Month 6
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 326 | 329
percentage of participants | 47.9 | 45.6
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; The analysis of RSDRL used a logistic regression (LREG) model, with country, sex, Baseline DRL, and treatment as fixed effects, and missing values were imputed using individual-patient predicted values of TAC derived from the MMRM model; Test type: Superiority or Other; p = 0.630, Adjusted Odds Ratio (OR) response; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.67 to 1.27]

4. Secondary Outcome: Change From Baseline in Clinical Status Using CGI-S
Description: The Clinical Global Impression - Severity of Illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline and Week 24
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 225 | 203
units on a scale | -1.04 (0.08) | -1.27 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; MMRM model with the Baseline score as a covariate, and site, sex, time in weeks, and treatment as fixed effects. The Baseline score-by-time and treatment-by-time interactions were also included in the model; an unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.029, Adjusted change from Baseline to Week 24; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.44 to -0.02], Standard Error of Mean 0.11 — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 225 participants in the placebo group and 203 participants in the nalmefene group

5. Secondary Outcome: Change in Clinical Status Using the CGI-I
Description: The Clinical Global Impression - Global Improvement (CGI-I) provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 24
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 225 | 203
units on a scale | 2.68 (0.08) | 2.51 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; MMRM model with the Baseline CGI-S score as a covariate, and site, sex, time in weeks, and treatment as fixed effects. The Baseline CGI-S score-by-time and treatment-by-time interactions were also included in the model. An unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.111, Adjusted change from Baseline to Week 24; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.38 to 0.04], Standard Error of Mean 0.11 — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Liver Function Test Gamma-glutamyl Transferase (GGT)
Description: GGT values
Time Frame: Week 24
Population: FAS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/L
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 224 | 207
IU/L | 44.9 (75.7) | 43.3 (75.2)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; Log-transformed GGT values were analysed using an MMRM model with the log-transformed Baseline value as a covariate, and site, sex, time in weeks, and treatment as fixed effects. Logtransformed Baseline value-by-time interaction and treatment-by-time interaction were included in the model. An unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.529, [Adjusted values; Ratio to placebo = 0.96, 95% CI 2-sided [0.86 to 1.08] — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 224 participants in the placebo group and 207 participants in the nalmefene group

7. Secondary Outcome: Liver Function Test Alanine Aminotransferase (ALAT)
Description: ALAT values
Time Frame: Week 24
Population: FAS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/L
Arm/Group | Placebo | Nalmefene 18.06 mg
Number analyzed (Participants) | 222 | 205
IU/L | 27.2 (56.3) | 25.0 (55.7)
Statistical Analysis 1: Comparison: Placebo vs Nalmefene 18.06 mg; Log-transformed ALAT values were analysed using an MMRM model with the log-transformed Baseline value as a covariate, and site, sex, time in weeks, and treatment as fixed effects. Logtransformed Baseline value-by-time and treatment-by-time interactions were included in the model. An unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.049, [Adjusted values; Ratio to placebo = 0.92, 95% CI 2-sided [0.84 to 1.00] — The Number of Participants Analyzed is participants with efficacy measurement available at this endpoint, that is, 222 participants in the placebo group and 205 participants in the nalmefene group

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 24 weeks, a 4-week run-out period, and a safety follow-up (visit/telephone call) scheduled for 4 weeks after completion of the study or after withdrawal from the study. Other Adverse Events: 24 weeks and a 4-week run-out period.
Arm/Group | Placebo | Nalmefene 18.06 mg
Serious Adverse Events (participants affected / at risk) | 14/337 | 7/341
Other Adverse Events (participants affected / at risk) | 102/337 | 157/341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=337) | Nalmefene 18.06 mg (N=341)
Myocardial infarction (Cardiac disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 3 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 2
Suicidal behaviour (Psychiatric disorders) | 1 | 0
Arteritis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=337) | Nalmefene 18.06 mg (N=341)
Diarrhoea (Gastrointestinal disorders) | 18 | 8
Nausea (Gastrointestinal disorders) | 20 | 59
Vomiting (Gastrointestinal disorders) | 8 | 19
Nasopharyngitis (Infections and infestations) | 20 | 22
Dizziness (Nervous system disorders) | 14 | 52
Headache (Nervous system disorders) | 26 | 43
Anxiety (Psychiatric disorders) | 17 | 11
Insomnia (Psychiatric disorders) | 23 | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The main publication has to be published before any sub publication. The investigators shall obtain Lundbeck's written approval before publishing any publication relating to nalmefene, the Study, the Protocol and/or the results recorded during the Study.